CLINICAL TRIAL: NCT01227889
Title: A Phase III Randomized, Open-label Study Comparing GSK2118436 to Dacarbazine (DTIC) in Previously Untreated Subjects With BRAF Mutation Positive Advanced (Stage III) or Metastatic (Stage IV) Melanoma
Brief Title: A Study Comparing GSK2118436 to Dacarbazine (DTIC) in Previously Untreated Subjects With BRAF Mutation Positive Advanced (Stage III) or Metastatic (Stage IV) Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113683
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-08

CONDITIONS: Cancer
Keywords: Metastatic melanoma; melanoma; BRAF mutant; Advanced melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — dabrafenib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GSK2118436 (Experimental): Subjects in this arm will receive GSK2118436 150 mg twice daily.
  Interventions: Drug: GSK2118436
- Dacarbazine (DTIC) (Active Comparator): Subjects will receive intravenous dacarbazine (DTIC) 1000 mg/m2 every 3 weeks
  Interventions: Drug: Dacarbazine (DTIC)
- Crossover (Experimental): Subjects who initially receive DTIC will be allowed to receive GSK2118436 after initial progression.
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — 150 mg twice daily
  Arms: Crossover; GSK2118436
Drug: Dacarbazine (DTIC) — Intravenous (IV), 1000 mg/m2 every 3 weeks until initial progression
  Arms: Dacarbazine (DTIC)

SUMMARY:
BRF113683 is a Phase III, randomized, open-label study comparing the efficacy, safety, and tolerability of GSK2118436 to dacarbazine (DTIC), in subjects with BRAF mutant advanced (Stage III) or metastatic (Stage IV) melanoma. Subjects will be randomized to receive 150 mg of GSK2118436 twice daily or 1000 mg/m2 DTIC every 3 weeks and continue on treatment until disease progression, death, or unacceptable adverse event. Subjects who progress on DTIC will be allowed to crossover to an optional extension arm of the study to receive GSK2118436.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Has advanced (unresectable Stage III) or metastatic (Stage IV) melanoma that is BRAF mutation positive (V600E)
* Is treatment naive for advanced (unresectable) or metastatic melanoma, with the exception of Interleukin 2 (IL-2) which is allowed.
* Has measurable disease according to RECIST 1.1 criteria.
* Women of child-bearing potential must have a negative pregnancy test within 14 days prior to the first dose of study treatment.
* Women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 4 weeks after the last dose of study medication.
* Men with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 16 weeks after the last dose of study medication.
* Must have adequate organ function.
* Must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy or surgery).
* Evidence of active central nervous system (CNS) disease.
* Previous treatment for metastatic melanoma, including treatment with BRAF or MEK inhibitor.
* A history of other malignancy. Subjects who have been disease-free for 5 years or subjects with a history of complete resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* History of Human Immunodeficiency Virus (HIV) infection.
* Certain cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2010-12-23 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (80):
- United States (11):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New York, New York
- Australia (4):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (4):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Villejuif
- Germany (21):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Jena, Thuringia
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
- Ireland (3):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
- Italy (8):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Terni, Umbria
  - GSK Investigational Site, Padua, Veneto
- GSK Investigational Site, Amsterdam, Netherlands
- Poland (5):
  - GSK Investigational Site, Brzozów
  - GSK Investigational Site, Konin
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Warsaw
- Russia (5):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
- Spain (6):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Hospitalet de Llobregat, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Seville

REFERENCES:
- [Background] Hauschild A, Grob JJ, Demidov LV, Jouary T, Gutzmer R, Millward M, Rutkowski P, Blank CU, Miller WH Jr, Kaempgen E, Martin-Algarra S, Karaszewska B, Mauch C, Chiarion-Sileni V, Martin AM, Swann S, Haney P, Mirakhur B, Guckert ME, Goodman V, Chapman PB. Dabrafenib in BRAF-mutated metastatic melanoma: a multicentre, open-label, phase 3 randomised controlled trial. Lancet. 2012 Jul 28;380(9839):358-65. doi: 10.1016/S0140-6736(12)60868-X. Epub 2012 Jun 25. PMID 22735384
- [Derived] Hauschild A, Ascierto PA, Schadendorf D, Grob JJ, Ribas A, Kiecker F, Dutriaux C, Demidov LV, Lebbe C, Rutkowski P, Blank CU, Gutzmer R, Millward M, Kefford R, Haas T, D'Amelio A Jr, Gasal E, Mookerjee B, Chapman PB. Long-term outcomes in patients with BRAF V600-mutant metastatic melanoma receiving dabrafenib monotherapy: Analysis from phase 2 and 3 clinical trials. Eur J Cancer. 2020 Jan;125:114-120. doi: 10.1016/j.ejca.2019.10.033. PMID 31864178
- [Derived] Santiago-Walker A, Gagnon R, Mazumdar J, Casey M, Long GV, Schadendorf D, Flaherty K, Kefford R, Hauschild A, Hwu P, Haney P, O'Hagan A, Carver J, Goodman V, Legos J, Martin AM. Correlation of BRAF Mutation Status in Circulating-Free DNA and Tumor and Association with Clinical Outcome across Four BRAFi and MEKi Clinical Trials. Clin Cancer Res. 2016 Feb 1;22(3):567-74. doi: 10.1158/1078-0432.CCR-15-0321. Epub 2015 Oct 7. PMID 26446943
- [Derived] Latimer NR, Abrams KR, Amonkar MM, Stapelkamp C, Swann RS. Adjusting for the Confounding Effects of Treatment Switching-The BREAK-3 Trial: Dabrafenib Versus Dacarbazine. Oncologist. 2015 Jul;20(7):798-805. doi: 10.1634/theoncologist.2014-0429. Epub 2015 Jun 3. PMID 26040620
- [Derived] Grob JJ, Amonkar MM, Martin-Algarra S, Demidov LV, Goodman V, Grotzinger K, Haney P, Kampgen E, Karaszewska B, Mauch C, Miller WH Jr, Millward M, Mirakhur B, Rutkowski P, Chiarion-Sileni V, Swann S, Hauschild A. Patient perception of the benefit of a BRAF inhibitor in metastatic melanoma: quality-of-life analyses of the BREAK-3 study comparing dabrafenib with dacarbazine. Ann Oncol. 2014 Jul;25(7):1428-1436. doi: 10.1093/annonc/mdu154. Epub 2014 Apr 25. PMID 24769640
- [Derived] Ouellet D, Gibiansky E, Leonowens C, O'Hagan A, Haney P, Switzky J, Goodman VL. Population pharmacokinetics of dabrafenib, a BRAF inhibitor: effect of dose, time, covariates, and relationship with its metabolites. J Clin Pharmacol. 2014 Jun;54(6):696-706. doi: 10.1002/jcph.263. Epub 2014 Jan 17. PMID 24408395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase III randomized, open-label study to compare GSK2118436 to Dacarbazine (DTIC) in previously untreated participants (par.) with BRAF mutation positive advanced (Stage III) or metastatic (Stage IV) melanoma. This study was conducted at 70 centers in 12 countries.
Pre-assignment Details: The study has 2 phases: Randomized and Crossover Phase. In Randomized Phase, a total of 250 par. were randomized in 3:1 to receive either oral dabrafenib 150 mg twice daily (BID) or intravenous DTIC 1000 milligram/meter square. Par. in DTIC arm with disease progression were considered for crossover to dabrafenib arm in Crossover Phase
Groups:
- GSK2118436 150 mg BID: Participants (par.) were randomly assigned to receive oral GSK2118436 150 milligrams (mg) twice a day (BID). Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until disease progression (DP), death, the occurrence of an unacceptable adverse event (AE), or withdrawal from the study. Participants who experienced investigator-reported DP but were benefitting from study treatment were permitted to continue GSK2118436 treatment upon approval of the GlaxoSmithKline Medical Monitor.
- DTIC 1000 mg/m^2 in RP; GSK2118436 in Crossover Phase: In the RP, par. received intravenous (IV) Dacarbazine (DTIC) 1000 mg per meters squared (mg/m^2) every 3 weeks. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Par. continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study. Par. who received DTIC in the RP and experienced DP had the option, at the discretion of the Investigator, of receiving GSK2118436 150 mg BID in the Crossover Phase. Par. who permanently discontinued DTIC treatment due to an AE, withdrawal of consent, or for any reason other than DP were not eligible for crossover to GSK2118436. Crossover par. continued on GSK2118436 until further DP was noted. After DP on GSK2118436, par. were followed for response, progression, survival, and further anti-cancer therapy.
Period: Randomized Phase (RP)
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP; GSK2118436 in Crossover Phase
Started | 187 | 63
Completed | 0 | 0
Not Completed | 187 | 63
Not completed — Adverse Event | 13 | 0
Not completed — Physician Decision | 13 | 5
Not completed — Progressive Disease | 135 | 52
Not completed — Study terminated by sponsor | 10 | 0
Not completed — Missing | 1 | 3
Not completed — Withdrawal by Subject | 15 | 3
Period: Crossover Phase
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP; GSK2118436 in Crossover Phase
Started | 0 | 37 (As of the data cut on December 18, 2012, 36 of 63 participants crossed over from DTIC to GSK2118436.)
Completed | 0 | 0
Not Completed | 0 | 37
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Progressive Disease | 0 | 31
Not completed — Study Terminated By Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK2118436 150 mg BID: Participants were randomly assigned to receive oral GSK2118436 150 mg BID. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study. Participants who experienced investigator-reported DP but were benefitting from study treatment were permitted to continue GSK2118436 treatment upon approval of the GlaxoSmithKline Medical Monitor.
- DTIC 1000 mg/m^2 in RP; GSK2118436 in Crossover Phase: In the RP, par. received IV DTIC 1000 mg/m^2 every 3 weeks. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Par. continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study. Par. who received DTIC in the RP and experienced DP had the option, at the discretion of the Investigator, of receiving GSK2118436 150 mg BID in the Crossover Phase. Par. who permanently discontinued DTIC treatment due to an AE, withdrawal of consent, or for any reason other than DP were not eligible for crossover to GSK2118436. Crossover par. continued on GSK2118436 until further DP was noted. After DP on GSK2118436, par. were followed for response, progression, survival, and further anti-cancer therapy.
- Total: Total of all reporting groups
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP; GSK2118436 in Crossover Phase | Total
Number analyzed (Participants) | 187 | 63 | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (13.76) | 51.6 (14.22) | 53.0 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 26 | 101
  Male | 112 | 37 | 149
Race/Ethnicity, Customized [Number; unit: participants]
  White | 186 | 63 | 249
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the interval of time between the date of randomization and the earlier of the date of disease progression or the date of death due to any cause. Disease progression was based on radiographic or photographic evidence, and assessments were made by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeters (mm). For participants who did not progress or die, PFS was censored at the date of last contact. Data are presented as median and 96% confidence interval.
Time Frame: Time interval between the date of randomization and the earlier of the date of disease progression or the date of death due to any cause (up to 9.9 months)
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not treatment was administered
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- GSK2118436 150 mg BID: Participants were randomly assigned to receive oral GSK2118436 150 milligrams (mg) twice a day (BID). Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until disease progression (DP), death, the occurrence of an unacceptable adverse event (AE), or withdrawal from the study. Participants who experienced investigator-reported DP but were benefitting from study treatment were permitted to continue GSK2118436 treatment upon approval of the GlaxoSmithKline Medical Monitor.
- DTIC 1000 mg/m^2 in RP: In the RP, participants received intravenous (IV) Dacarbazine (DTIC) 1000 milligrams per meters squared (mg/m^2) every 3 weeks. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 63
Months | 6.9 [5.5 to 9.0] | 2.7 [1.4 to 3.2]
Statistical Analysis 1: Comparison: GSK2118436 150 mg BID vs DTIC 1000 mg/m^2 in RP; Test type: Superiority or Other; p < 0.0001, Log Rank — The p value from a stratified log-rank test was adjusted for disease stage at screening; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.26 to 0.60] — HRs were estimated using a Pike estimator. HR from a stratified log-rank test was adjusted for disease stage at screening

2. Primary Outcome: Progression-free Survival (PFS) as Assessed by an Independent Radiologist: Randomized Phase
Description: PFS is defined as the interval of time between the date of randomization and the earlier of the date of disease progression or the date of death due to any cause. Disease progression was based on radiographic or photographic evidence, and assessments were made by an independent radiologist according to RECIST version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. For participants who did not progress or die, PFS was censored at the date of last contact.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- DTIC 1000 mg/m^2 in RP: In the RP, participants received IV DTIC 1000 mg/m^2 every 3 weeks. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 63
Months | 6.7 [5.0 to 6.9] | 2.9 [1.7 to 4.9]
Statistical Analysis 1: Comparison: GSK2118436 150 mg BID vs DTIC 1000 mg/m^2 in RP; Test type: Superiority or Other; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.20 to 0.61] — HRs were estimated using a Pike estimator. HR was adjusted for disease stage at screening

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval of time between the date of randomization and the date of death due to any cause. For participants who did not die, overall survival was censored at the date of last contact.
Time Frame: Time interval between the date of randomization and the date of death due to any cause (up to 22.1 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- DTIC 1000 mg/m^2 in RP: In the RP, participants received IV DTIC 1000 mg/m^2 every 3 weeks. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants. continued on treatment until DP, death, the occurrence of an unacceptable AE, or withdrawal from the study.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 63
Months | 20.0 [16.7 to 24.2] | 15.6 [11.9 to 21.2]
Statistical Analysis 1: Comparison: GSK2118436 150 mg BID vs DTIC 1000 mg/m^2 in RP; Test type: Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.57 to 1.18] — HRs were estimated using a Pike estimator. HR was adjusted for disease stage at screening

4. Secondary Outcome: Number of Participants With a Best Overall Response of Confirmed Complete Response (CR) or Confirmed Partial Response (PR) as Assessed by the Investigator: Randomized Phase
Description: A participant was defined as a responder if he/she achieved either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Response was evaluated by an investigator per RECIST, version 1.1. A participant without a post-Baseline assessment of response was considered a non-responder. Confirmation, per RECIST version 1.1, requires a confimatory disease assessment of CR or PR at least 28 days after the initial disease assessment of CR or PR.
Time Frame: From randomization until the first documented evidence of a confirmed complete response or partial response (median of 6.6 weeks)
Population: ITT Population
Measure: Number; unit: participants
Groups:
- GSK2118436 150 mg BID: Participants were randomly assigned to receive oral GSK2118436 150 mg BID. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until disease DP, death, the occurrence of an unacceptable adverse AE, or withdrawal from the study. Participants who experienced investigator-reported DP but were benefitting from study treatment were permitted to continue GSK2118436 treatment upon approval of the GlaxoSmithKline Medical Monitor.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 63
participants
  CR | 26 | 4
  PR | 86 | 11

5. Secondary Outcome: Number of Participants With a Best Overall Response of Confirmed CR or PR as Assessed by an Independent Radiologist: Randomized Phase
Description: A participant was defined as a responder if he/she achieved either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Response was evaluated by an independent radiologist per RECIST, version 1.1. A participant without a post-Baseline assessment of response was considered a non-responder. Confirmation, per RECIST version 1.1, requires a confimatory disease assessment of CR or PR at least 28 days after the initial disease assessment of CR or PR.
Time Frame: From randomization until the first documented evidence of a confirmed complete response or partial response (median of 12.0 weeks)
Population: ITT Population
Measure: Number; unit: participants
Groups:
- GSK2118436 150 mg BID: Participants were randomly assigned to receive oral GSK2118436 150 mg BID. Dose reductions were permitted based on the severity of the hematological toxicity. Stopping recommendations for study treatment were also provided for cases of reoccurring skin toxicity, cardiovascular complication or abnormalities, and liver abnormalities. Participants continued on treatment until disease DP, death, the occurrence of an unacceptable AE, or withdrawal from the study. Participants who experienced investigator-reported DP but were benefitting from study treatment were permitted to continue GSK2118436 treatment upon approval of the GlaxoSmithKline Medical Monitor.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 63
participants
  CR | 6 | 1
  PR | 87 | 3

6. Secondary Outcome: Duration of Response as Assessed by the Investigator: Randomized Phase
Description: Duration of response for participants with either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) was defined as the time from the first documented evidence of a PR or CR until the first documented sign of PD or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: Time from the first documented evidence of PR or CR until the first documented sign of disease progression or death due to any cause (up to 65.6 weeks)
Population: ITT Population. Only participants with a confirmed CR or PR were assessed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 112 | 15
Months | 9.2 [7.4 to 11.9] | 8.2 [3.5 to 18.3]

7. Secondary Outcome: Duration of Response as Assessed by an Independent Radiologist: Randomized Phase
Description: Duration of response for participants with either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) was defined as the time from the first documented evidence of a PR or CR until the first documented sign of PD or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. NA indicates that data is not available.
Time Frame: Time from the first documented evidence of PR or CR until the first documented sign of disease progression or death due to any cause (up to 7.4 months)
Population: ITT Population. Only participants with a confirmed CR or PR were assessed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 93 | 4
Months | 5.5 [5.0 to 6.7] | NA [NA to NA] — Median duration of response could not be calculated because there were not enough participants with a CR or PR.

8. Secondary Outcome: Progression-free Survival (PFS2) as Assessed by the Investigator: Crossover Phase
Description: PFS2 is defined as the time from the first dose of GSK2118436, in participants randomized to DTIC who crossed over to GSK2118436 after initial progression, to the earliest date of radiographic or photographic disease progression or death due to any cause. Disease progression was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. For participants who did not progress or die, PFS was censored at the date of last contact.
Time Frame: Time from first dose of GSK2118436 in participants who crossover after initial progression to the earliest date of radiographical or photographical PD or death due to any cause (up to 6.4 months)
Population: Crossover Treatment Population: the subset of participants who were randomized to the DTIC arm, and who elected at the point of disease progression to receive GSK2118436. Only participants who received at least one dose of GSK2118436 were included in the Crossover Treatment Population.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- GSK25118436 in Crossover Phase: Participants who received DTIC in the RP and experienced DP had the option, at the discretion of the Investigator, of receiving GSK2118436 150 mg BID in the Crossover Phase. Participants who permanently discontinued DTIC treatment due to an AE, withdrawal of consent, or for any reason other than DP were not eligible for crossover to GSK2118436. Crossover participants continued on GSK2118436 until further DP was noted. After DP on GSK2118436, participants were followed for response, progression, survival, and further anti-cancer therapy.
Arm/Group | GSK25118436 in Crossover Phase
Number analyzed (Participants) | 37
Months | 4.3 [4.1 to 6.1]

9. Secondary Outcome: Number of Participants With a Best Overall Response of Confirmed Complete Response (CR) or Confirmed Partial Response (PR) as Assessed by the Investigator: Crossover Phase
Description: as for outcome 4
Time Frame: From randomization until the first documented evidence of a confirmed complete response or partial response (up to 6.4 months)
Population: Crossover Treatment Population. At the time data were analyzed for overall response, only 37 participants had crossed over from DTIC treatment to GSK25118436 treatment.
Measure: Number; unit: participants
Arm/Group | GSK25118436 in Crossover Phase
Number analyzed (Participants) | 37
participants
  CR | 0
  PR | 12

10. Secondary Outcome: Duration of Response as Assessed by the Investigator: Crossover Phase
Description: as for outcome 6
Time Frame: Time from the first documented evidence of PR or CR until the first documented sign of disease progression or death due to any cause (up to 6.4 months)
Population: Crossover Population. Only participants with a confirmed CR or PR were assessed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK25118436 in Crossover Phase
Number analyzed (Participants) | 12
Months | 4.4 [2.5 to 6.2]

11. Secondary Outcome: Number of Participants With Non-melanoma Skin Lesions: Randomized Phase
Description: Dermatological examinations were performed by the investigator, or at the discretion of the investigator, referred to a dermatologist. The number of participants with non-melanoma skin lessions was assessed from the time of Screening until study completion or discontinuation from the study for any reason.
Time Frame: From Screening until study completion or discontinuation from the study (up to 9.9 months)
Population: Safety Population: all randomized participants who received at least one dose of study drug, based on the actual treatment received, if this differed from that to which the participant was randomized
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP
Number analyzed (Participants) | 187 | 59
participants
  Number of Subjects with Event | 14 | 0
  Number of Events | 24 | 0

12. Secondary Outcome: Agreement Rate for V600E Mutation Validation of the BRAF Mutation Assay
Description: Analytical and clinical validation of the companion diagnostic (cDx) assay was performed to determine the extent of agreement between the bioMerieux cDx assay (THxID BRAF Assay) and the Clinical Trial Assay (CTA) to detect BRAF mutations to determine participant eligibility into the study. Skin tissue samples collected at the Screening visit were used for this analysis. Multiple specimen per participant were analyzed.
Time Frame: Screening
Population: V600E positive participants screened for BREAK-3 study
Measure: Number (95% Confidence Interval); unit: Percent agreement
Groups:
- All Screened Participants: Specimens were tested for V600E mutations to determine trial eligibility with the CTA were retested with the THxID BRAF test. The analytical agreement between the THxID BRAF and the CTA was evaluated for both mutation positive and mutation negative specimens from all sites.
Arm/Group | All Screened Participants
Number analyzed (Participants) | 734
Percent agreement
  Agreement for V600E | 96.70 [93.6 to 98.3]
  Agreement for V600K | 90.00 [78.6 to 95.7]
  Agreement for mutation negative | 95.00 [91.6 to 97.0]
  Agreement for overall | 94.90 [92.7 to 96.4]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product to the end of the study. The total duration of the study including a long-term follow-up phase was up to 5 years.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of study drug, based on the actual treatment received, if this differed from that to which the participant was randomized.
Groups:
- GSK25118436 in the Crossover Phase: Participants who received DTIC in the RP and experienced DP had the option, at the discretion of the Investigator, of receiving GSK2118436 150 mg BID in the Crossover Phase. Participants who permanently discontinued DTIC treatment due to an AE, withdrawal of consent, or for any reason other than DP were not eligible for crossover to GSK2118436. Crossover participants continued on GSK2118436 until further DP was noted. After DP on GSK2118436, participants were followed for response, progression, survival, and further anti-cancer therapy.
Arm/Group | GSK2118436 150 mg BID | DTIC 1000 mg/m^2 in RP | GSK25118436 in the Crossover Phase
All-Cause Mortality (participants affected / at risk) | 5/187 | 0/59 | 1/37
Serious Adverse Events (participants affected / at risk) | 64/187 | 14/59 | 9/37
Other Adverse Events (participants affected / at risk) | 181/187 | 51/59 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2118436 150 mg BID (N=187) | DTIC 1000 mg/m^2 in RP (N=59) | GSK25118436 in the Crossover Phase (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (4) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 10 (13) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 3 (5) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (11) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (12) | 0 (0) | 2 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2118436 150 mg BID (N=187) | DTIC 1000 mg/m^2 in RP (N=59) | GSK25118436 in the Crossover Phase (N=37)
Anaemia (Blood and lymphatic system disorders) | 10 (14) | 7 (9) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 10 (18) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 8 (11) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (16) | 7 (8) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 11 (20) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 27 (32) | 8 (9) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 31 (42) | 7 (8) | 4 (5)
Nausea (Gastrointestinal disorders) | 55 (69) | 29 (49) | 9 (9)
Vomiting (Gastrointestinal disorders) | 42 (55) | 15 (19) | 5 (5)
Asthenia (General disorders) | 37 (56) | 9 (11) | 6 (8)
Chills (General disorders) | 23 (40) | 0 (0) | 4 (5)
Fatigue (General disorders) | 48 (57) | 14 (21) | 6 (6)
Influenza like illness (General disorders) | 14 (16) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 12 (13) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 61 (102) | 8 (8) | 9 (11)
Folliculitis (Infections and infestations) | 11 (13) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 35 (57) | 4 (6) | 4 (8)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (13) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (7) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 4 (5) | 0 (0)
Weight decreased (Investigations) | 13 (13) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 3 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 26 (34) | 6 (7) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (19) | 3 (4) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 11 (13) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 74 (111) | 0 (0) | 16 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (48) | 4 (4) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 (20) | 0 (0) | 6 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (41) | 0 (0) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (40) | 6 (7) | 6 (6)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (20) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (18) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (23) | 0 (0) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (55) | 0 (0) | 3 (3)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 (85) | 0 (0) | 10 (15)
Dizziness (Nervous system disorders) | 15 (17) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 68 (109) | 5 (6) | 6 (7)
Paraesthesia (Nervous system disorders) | 12 (13) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 10 (10) | 5 (5) | 3 (3)
Insomnia (Psychiatric disorders) | 16 (19) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (42) | 4 (6) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 22 (51) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 54 (59) | 0 (0) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 28 (36) | 0 (0) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 18 (28) | 0 (0) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 13 (14) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 71 (156) | 0 (0) | 11 (20)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 (44) | 0 (0) | 5 (5)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 17 (20) | 0 (0) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 35 (45) | 0 (0) | 10 (13)
Skin lesion (Skin and subcutaneous tissue disorders) | 14 (18) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 10 (16) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 2 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (4)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (5)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.